CLINICAL TRIAL: NCT05892081
Title: Effect of Colloidal Oatmeal Compared to Colloid Cream on Diaper Rash Among Preterm Neonates in the Neonatal Intensive Care Unit.
Brief Title: Colloidal Oatmeal, Colloid Cream, Diaper Rash, Preterm Neonates and Neonatal Intensive Care Unit
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seham El-Sayed Saleh Hassan (Other)
Responsible Party: Sponsor-Investigator, Seham El-Sayed Saleh Hassan, Lecturer of pediatric nursing, faculty of nursing, Matrouh University
Organization: Matrouh University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Document attached-Not given
Record Dates: First submitted 2023-04-11; First posted 2023-06-07 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Diaper Rash; Preterm Neonates
Keywords: Colloidal oatmeal; Diaper rash; Preterm neonates
MeSH Terms: conditions — Diaper Rash

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (No Intervention): The control group received the usual care of the unit.
- Colloid group (Experimental): Received cold cream three times a day on the rash area while diaper changing by the researcher plus the usual care
  Interventions: Biological: Cold cream
- Colloid oatmeal group (Experimental): Received colloid oatmeal cream three times a day on the rash area while diaper changing by the researcher plus the usual care
  Interventions: Biological: Colloidal oatmeal

INTERVENTIONS:
Biological: Colloidal oatmeal — The colloid oatmeal had the following component: Colloidal Oat (5gm), stearic acid 5, cretoctryl alcohol 2.5, cetyl alcohol 2.5, koh 02, potassium sorbate 1gm, paraffin oil 5ml, and soft paraffin 10gm
  Arms: Colloid oatmeal group
Biological: Cold cream — It is composed of stearic acid 5, cretoctryl alcohol 2.5, cetyl alcohol 2.5, koh 02, potassium sorbate 1gm, paraffin oil 5ml, and soft paraffin 10gm
  Arms: Colloid group

SUMMARY:
-This study aimed to investigate the effect of colloid oatmeal compared to colloid cream on diaper rash among preterm neonates in the NICU.

DETAILED DESCRIPTION:
A quasi-experimental study was carried out in the NICU of El-Raml Children's Hospital at Wengat in Alexandria. Ninety preterm neonates were randomly assigned to three equal groups. The control group received the usual care of NICU for diaper rash, colloidal oatmeal group received colloidal oatmeal cream and colloid group received colloid cream (cold which is the base for colloid oatmeal)

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates
* Have diaper rash,
* Hemodynamically stable
* Receive enteral feeding (breast, bottle, gavage, or mixed feeding)
* Newly admitted to the previously mentioned setting
* On the first day of exposure to diaper rash

Exclusion Criteria:

* Preterm who have candida infection in groin
* Use other drugs for diaper rash

Ages: 34 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Preterm neonates who receive colloid assessed by rash scale score. | four days
  Mild degree of diaper rash score will mean improvement in diaper rash

CONTACTS AND LOCATIONS:
Locations (1):
- Matrouh university, Marsá Maţrūḩ, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Academy of Pediatrics. (2014). Diaper rash. Available from: http//www.pdf secret.com _diaper-rash-southwest-childrens-center.pdf.
- [Background] Altmann T, Fischman. (2018). The dreaded diaper rash: A pediatrician's advice for preventing and treating an angry bottom. The dreaded diaper rash: A pediatrician's advice for preventing and treating an angry bottom - The Washington Post.
- [Background] Association of Women's Health, Obstetric and Neonatal Nurses (AWHONN). Neonatal skin care evidence-based clinical practice guideline (3rd ed.). Washington, DC; (2013).
- [Background] Baudouin C, Lachmann N, Rocheteau J, Chadoutaud B, Boy E, Leclere-Bienfait S. Diaper dermatitis management: a global and innovative strategy for a new generation of skin care. J Am Acad Dermatol, 2015; 72(5):199.
- [Background] Blume-Peytavi U, Lavender T, Jenerowicz D, Ryumina I, Stalder JF, Torrelo A, Cork MJ. Recommendations from a European Roundtable Meeting on Best Practice Healthy Infant Skin Care. Pediatr Dermatol. 2016 May;33(3):311-21. doi: 10.1111/pde.12819. Epub 2016 Feb 26. PMID 26919683
- [Background] Blume-Peytavi U, Hauser M, Lunnemann L, Stamatas GN, Kottner J, Garcia Bartels N. Prevention of diaper dermatitis in infants--a literature review. Pediatr Dermatol. 2014 Jul-Aug;31(4):413-29. doi: 10.1111/pde.12348. Epub 2014 May 29. PMID 24890321
- [Background] Boyles, M. (2022).Health Benefits of Oatmeal and Oats. Available from: http//.www.Health Benefits of Oatmeal & Oats | Oatmeal to Soothe Itchy Skin | The Old Farmer's Almanac.
- [Background] Buckley BS, Mantaring JB, Dofitas RB, Lapitan MC, Monteagudo A. A New Scale for Assessing the Severity of Uncomplicated Diaper Dermatitis in Infants: Development and Validation. Pediatr Dermatol. 2016 Nov;33(6):632-639. doi: 10.1111/pde.12988. Epub 2016 Sep 22. PMID 27653955
- [Background] Burdall O, Willgress L, Goad N. Neonatal skin care: Developments in care to maintain neonatal barrier function and prevention of diaper dermatitis. Pediatr Dermatol. 2019 Jan;36(1):31-35. doi: 10.1111/pde.13714. Epub 2018 Dec 2. PMID 30506880
- [Background] Chat, S., Uppal, S., Kearns, D., Ashin, J. Colloidal Oatmeal in the Treatment of Atopic Dermatitis Is this plant-based intervention an effective treatment alternative? By Practical Dermatology. 2020.
- [Background] Collier M, Simon D. Protecting vulnerable skin from moisture-associated skin damage. Br J Nurs. 2016 Nov 10;25(20 Suppl):S26-S32. doi: 10.12968/bjon.2016.25.20.S26. PMID 27834525
- [Background] Furber C, Bedwell C, Campbell M, Cork M, Jones C, Rowland L, Lavender T. The challenges and realties of diaper area cleansing for parents. J Obstet Gynecol Neonatal Nurs. 2012 Nov-Dec;41(6):E13-25. doi: 10.1111/j.1552-6909.2012.01390.x. Epub 2012 Jul 23. PMID 22822929
- [Background] Gregorio J, and Rodriguez K. Diaper Dermatitis in Infant Skin: Causes and Mitigation. neonatal INTENSIVE CARE. 2017; 30 (3):38-40.
- [Background] Hugill K. Revisiting infant nappy dermatitis: causes and preventive care. Br J Midwifery, 2017;25(3):150-54.
- [Background] Ilnytska O, Kaur S, Chon S, Reynertson KA, Nebus J, Garay M, Mahmood K, Southall MD. Colloidal Oatmeal <em>(Avena Sativa)</em> Improves Skin Barrier Through Multi-Therapy Activity. J Drugs Dermatol. 2016 Jun 1;15(6):684-90. PMID 27272074
- [Background] Klunk C, Domingues E, Wiss K. An update on diaper dermatitis. Clin Dermatol. 2014 Jul-Aug;32(4):477-87. doi: 10.1016/j.clindermatol.2014.02.003. Epub 2014 Feb 28. PMID 25017459
- [Background] Madhu R, Vijayabhaskar C, Anandan V, Nedunchelian K, Thangavelu S, Soans ST, Shastri DD, Parekh BJ, Kumar RR, Basavaraja GV. Indian Academy of Pediatrics Guidelines for Pediatric Skin Care. Indian Pediatr. 2021 Feb 15;58(2):153-161. PMID 33632947
- [Background] Merrill L. Prevention, Treatment and Parent Education for Diaper Dermatitis. Nurs Womens Health. 2015 Aug-Sep;19(4):324-36; quiz 337. doi: 10.1111/1751-486X.12218. PMID 26264797
- [Background] Morris H. The bottom line on nappy rash. Br J Midwifery, 2012; 20 (9):623-26.
- [Background] Narayanan V, Ganjoo A, Kadhe G. Efficacy and Tolerability of an Oatmeal Moisturizer Containing Colloidal Oatmeal for Dry Skin Conditions: A Post-marketing Study. Indian Journal of Clinical Practice. 2016; 27(1): 1118-23.
- [Background] Paller A , Mancini A. Hurwitz Clinical Pediatric Dermatology: A Textbook of Skin Disorders of Childhood and Adolescence. 6thEd. Elsevier Saunders, 2011.
- [Background] Panahi Y, Sharif MR, Sharif A, Beiraghdar F, Zahiri Z, Amirchoopani G, Marzony ET, Sahebkar A. A randomized comparative trial on the therapeutic efficacy of topical aloe vera and Calendula officinalis on diaper dermatitis in children. ScientificWorldJournal. 2012;2012:810234. doi: 10.1100/2012/810234. Epub 2012 Apr 19. PMID 22606064
- [Background] Pazyar N, Yaghoobi R, Kazerouni A, Feily A. Oatmeal in dermatology: a brief review. Indian J Dermatol Venereol Leprol. 2012 Mar-Apr;78(2):142-5. doi: 10.4103/0378-6323.93629. PMID 22421643
- [Background] Sarin, A., Bhatia, J., Sarkar, R.. Diaper Dermatitis. Asian Journal of Pediatric Dermatology AJPD. 2021; 4 (1): 2.